CLINICAL TRIAL: NCT03318822
Title: Usability and Tolerability of Novel Protection Device Against Potential Brain Injury During Competitive Sport
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Greg Myer, Associate Professor, Emory University
Other Study IDs: STUDY00001960; 2016-9625 (Other: CCHMC)
Record Dates: First submitted 2017-08-21; First posted 2017-10-24 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Brain Injuries, Traumatic; Brain Injury Traumatic Mild
Keywords: brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Q-Collar: Subjects wearing the Q-Collar
  Interventions: Device: Q-Collar

INTERVENTIONS:
Device: Q-Collar — An externally-worn medical device that applies mild jugular compression

SUMMARY:
The purpose of the study is to assess the usability and tolerability of this jugular vein compression device in a population of helmeted and non-helmeted competitive high school, collegiate and professional athletes in the sports of football and rugby. This study differs from previous work in that it is designed to capture additional data related to the athlete experience wearing the jugular vein compression device in older and more elite playing levels.

DETAILED DESCRIPTION:
Significant morbidity, mortality, and related costs are caused by traumatic brain injury (TBI). A simple, effective, and lightweight device worn by athletes or war fighters in the field, designed to mitigate TBI resulting from blast trauma or concussive events, would save lives, and the huge costs incurred for life-treatment of surviving victims. An externally-worn medical device that applies mild jugular compression according to the principle of the Queckenstedt Maneuver (the Device) is being developed by Q30 Sports Science, LLC (Q30). Preliminary research suggests that the Device has the potential to reduce the likelihood of TBI. The currently developed collar has been approved for studies in humans and the results indicate safety for use during high demand and maximal exertion activities. Regarding safety, the externally worn collar is meticulously designed to mimic the body's own omohyoid muscle actions upon the jugular veins that will provide similar pressure and volume increases not to surpass that of a yawn or the mere act of just lying down. This study will investigate the tolerability of this device in athletes participating in the competitive sports of football and rugby at the high school, collegiate or professional levels.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteer
* Able to provide written consent
* Must be 14 years or older and a participant in collegiate/professional sports of football or rugby

Exclusion Criteria:

* Unable to provide written consent
* History of neurological deficits, previous cerebral infarction, or severe head trauma as indicated through pre-season screening:
* Medical contraindications to restriction of venous outflow via the internal jugular veins (known increased intracerebral pressure, metabolic acidosis or alkalosis)
* Glaucoma (Narrow Angle or Normal Tension)
* Hydrocephalus
* Recent penetrating brain trauma (within 6 months)
* Known carotid hypersensitivity
* Known increased intracranial pressure
* Central vein thrombosis
* Any known airway obstruction
* Any known seizure disorder

Ages: 14 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Normal healthy volunteers aged 14-49
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Tolerability of collar usage | 1 year
  measure subject tolerability to wearing the device via weekly survey

SECONDARY OUTCOMES:
Compliance of collar usage | 1 year
  measure subject compliance to wearing the device via weekly survey completion

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Cincinnati Childrens Hospital
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No